CLINICAL TRIAL: NCT05905952
Title: Evaluation of Postural Stability and Ankle Mobility in Haglund Syndrome
Brief Title: Postural Stability and Ankle Mobility in Haglund Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nassif Magdy Mousa, principle investigator, Cairo University
Other Study IDs: P.T.REC/ 012/004497
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Haglund Deformity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: to twenty five patient of Haglund syndrome as (patient group) after being diagnosed and referred by orthopedic surgeon and twenty
  Interventions: Diagnostic Test: balance and ROM assessment
- control group: twenty five Healthy volunteers as (control group) based on the following inclusion and exclusion criteria
  Interventions: Diagnostic Test: balance and ROM assessment

INTERVENTIONS:
Diagnostic Test: balance and ROM assessment — assessment of postural stability and ankle range of motion

SUMMARY:
The purpose of the study is to find out the impact of Haglund syndrome on ankle plantarflexion and dorsiflexion ROM, dynamic postural stability and fall risk.

DETAILED DESCRIPTION:
This study will be delimited to:

* Total sample size is fifty participants, twenty five patient of symptomatic Haglund syndrome of both gender and twenty five healthy volunteers of matched age, sex and body mass index without any musculoskeletal complaints of the lower limbs.
* Biodex balance system will be used to determine postural stability.
* Ankle plantarflexion and dorsiflexion range of motion will be measured using an Electrogoniometer.
* Age of the patients 25-56
* BMI of (18.5 to 24.9)

Participants:

Fifty volunteers from both genders will participate in the study. They will be assigned from outpatient clinic of Faculty of Physical Therapy, Deraya University. They will be interviewed and divided to twenty five patient of Haglund syndrome as (patient group) after being diagnosed and referred by orthopedic surgeon and twenty five Healthy volunteers as (control group) based on the following inclusion and exclusion criteria:

ELIGIBILITY:
Inclusion Criteria:

* For patient group:

  * Patient referred from orthopedic surgeon with diagnoses as Haglund syndrome according to the following signs and symptoms
  * Calcaneal prominence diagnosed on lateral weight bearing radiograph with bony prominence superior to parallel pitch lines or posterior calcaneal angle greater than 75 degrees
  * Pain medially at insertion of tendo-achilles
  * Palpation of hard, bony prominence
  * Pain upon rising out of bed
  * Both unilateral and bilateral cases, and in consideration of dealing with bilateral cases the tested limb will be the most painful limb.
  * Age of 25-56 years
  * Both males and females.
  * BMI of (18.5 to 24.9)

For control group:

Healthy volunteers of matched age, sex and body mass index without any musculoskeletal complaints of the lower limbs and will be included in the control group in this study .

Exclusion Criteria:

* Musculoskeletal disorders except Haglund syndrome
* cognitive disorder, visual impairment that affected their daily living and any further medical condition that would prohibit them from participating safely in the chosen balance measures
* sensory loss at foot or ankle and with a systemic inﬂammatory disease, such as diabetes mellitus, peripheral neuropathy, rheumatoid arthritis and ankylosing spondylitis, who had undergone corticosteroid injections or physical therapy in the last three months
* Patients with vestibular or neurological disorders
* Any other cause of posterior heel pain.

Ages: 25 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with Haglund syndrome
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
postural stability test report | 1 day
  a measurement of the antero-posterior, medio-lateral and overall stability and range of motion
ankle range of motion test | 1 day
  measuring of ankle planter and dorsiflexion range of motion with digital goniometer

CONTACTS AND LOCATIONS:
Overall Officials: enas F youssif, prof, Principal Investigator — Cairo University
Locations (1):
- Deraya University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publication in peer-reviewed journals
Supporting Information: Study Protocol, SAP
Time Frame: year